CLINICAL TRIAL: NCT03441971
Title: Evaluation of the GORE PV1 Device for Replacement of the Pulmonary Valve and Reconstruction of Right Ventricular Outflow Tract
Brief Title: Evaluation of the GORE PV1 Device in Patients With Pulmonary Valve Dysfunction
Status: Active, not recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: W.L.Gore & Associates (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Device Feasibility
Other Study IDs: Gore PVC 17-02
Record Dates: First submitted 2018-02-15; First posted 2018-02-22 (Actual); Last update posted 2026-02-05 (Actual); Status verified 2026-02

CONDITIONS: Heart Defects, Congenital; Tetralogy of Fallot; Pulmonary Valve Insufficiency; Pulmonary Valve Stenosis
MeSH Terms: conditions — Heart Defects, Congenital; Tetralogy of Fallot; Pulmonary Valve Insufficiency; Pulmonary Valve Stenosis

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: Yes | Unapproved Device: Yes

ARMS (1):
- Single Arm (Experimental): Participants will receive the device on Day 1.
  Interventions: Device: GORE PV1

INTERVENTIONS:
Device: GORE PV1 — Implantation of GORE PV1 Device for procedure to replace the pulmonary valve and reconstruct the right ventricular outflow tract (RVOT).

SUMMARY:
This study will assess the safety and performance of the GORE PV1 Device for replacement of the pulmonary valve and reconstruction of the Right Ventricular Outflow Tract (RVOT).

ELIGIBILITY:
Inclusion Criteria:

1. A symptomatic or appropriate asymptomatic subject with a native or repaired right ventricular outflow tract requiring reconstruction with a valved conduit
2. Age ≥5 years at the time of informed consent signature.

Note: Additional Inclusion Criteria may apply

Exclusion Criteria:

1. An artificial valve at another position or will need an artificial valve at another position (i.e. replacement at the time of index procedure or anticipated within 3 years).
2. Subjects with previously implanted pacemaker (including defibrillators).
3. Major or progressive non-cardiac disease (liver failure, renal failure, cancer) that has a life expectancy of less than one year.

Note: Additional Exclusion Criteria may apply

Min Age: 5 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 15 (Estimated)
Dates: Start 2018-06-07 (Actual); Primary Completion 2020-04-13 (Actual); Study Completion 2030-03 (Estimated)

PRIMARY OUTCOMES:
Valve-related mortality and device-related re-intervention | 6 months
  The composite of valve-related mortality and device-related re-intervention measured at 6 months post-procedure

SECONDARY OUTCOMES:
MRI change in right ventricular end diastolic volume index | 6 months
  Six month change from baseline in right ventricular end diastolic volume index as measured from Magnetic Resonance Imaging
MRI change in right ventricular end systolic volume index at 6 months | 6 months
  Six month change from baseline in right ventricular end systolic volume index as measured from Magnetic Resonance Imaging
MRI change in left ventricular diastolic volume index at 6 months | 6 months
  Six month change from baseline in left ventricular diastolic volume index as measured from Magnetic Resonance Imaging
MRI change in right ventricular ejection fraction at 6 months | 6 months
  Six month change from baseline in right ventricular ejection fraction index as measured from Magnetic Resonance Imaging
Echo change in right ventricular diastolic area at 12 months | 12 months
  Twelve month change from baseline in right ventricular diastolic area as measured from echocardiography
Echo change in right ventricular systolic area at 12 months | 12 months
  Twelve month change from baseline in right ventricular systolic area as measured from echocardiography
Echo change in left ventricular end diastolic volume index at 12 months | 12 months
  Twelve month change from baseline in left ventricular end diastolic volume index as measured from echocardiography
Echo change in right ventricular fractional area change at 12 months | 12 months
  Twelve month change from baseline in right ventricular fractional area change as measured from echocardiography
Six month mean pressure gradient <= 40 mmHG | 6 months
  Number of subjects with mean pressure gradient across conduit (RV to PA) less than or equal to 40 mmHg at 6 months
Twelve month mean pressure gradient <= 40 mmHG | 12 months
  Number of subjects with mean pressure gradient across conduit (RV to PA) less than or equal to 40 mmHg at 12 months
Six month pulmonary regurgitation < moderate | 6 months
  Number of subjects with pulmonary regurgitation less than moderate at 6 months
Twelve month pulmonary regurgitation < moderate | 12 months
  Number of subjects with pulmonary regurgitation less than moderate at 12 months
Device-related re-intervention at 1, 3, 6, 12, 24, 36, 48, and 60 months | 1, 3, 6, 12, 24, 36, 48, and 60 months
  Kaplan-Meier estimates of device-related re-intervention summarized at 1, 3, 6, 12 months, and annually through 5 years
All-cause mortality at 1, 3, 6, 12, 24, 36, 48, and 60 months | 1, 3, 6, 12, 24, 36, 48, and 60 months
  Kaplan-Meier estimates of all-cause mortality summarized at 1, 3, 6, 12 months, and annually through 5 years

CONTACTS AND LOCATIONS:
Overall Officials: Pedro del Nido, MD, Principal Investigator — Boston Children's Hospital
Locations (3):
- United States (3):
  - Lurie Children's Hospital, Chicago, Illinois
  - Boston Children's Hospital, Boston, Massachusetts
  - Nationwide Children's Hospital, Columbus, Ohio

IPD SHARING:
Plan to Share IPD: No